CLINICAL TRIAL: NCT00260169
Title: Patient-Centered Depression Care in the Public Sector
Brief Title: Determining Depression Treatment Preferences of Low-Income Latinos in Primary Care Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Isabel T. Lagomasino, MD, MSHS, Study Principal Investigator, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH067949 (NIH); R01MH067949 (NIH); DSIR 82-SEPC
Record Dates: First submitted 2005-11-29; First posted 2005-12-01 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Depression
Keywords: Treatment Preferences; Public sector; Latino
MeSH Terms: conditions — Depression

ARMS (2):
- 1 (Experimental): Participants will receive collaborative care
  Interventions: Behavioral: Collaborative care treatment
- 2 (Active Comparator): Participants will receive enhanced usual care
  Interventions: Behavioral: Enhanced usual care

INTERVENTIONS:
Behavioral: Collaborative care treatment — Patients receiving collaborative care treatment choose 12 weeks of CBT and/or medication management (antidepressants prescribed by patients' primary care provider) from the study depression care specialist (DCS).
  Arms: 1
Behavioral: Enhanced usual care — Usual care participants are assigned to a 16-week wait-list for the study treatment, during which they are free to receive treatment elsewhere. A letter is given to participants' primary care providers (PCP) that indicates they screened positive for depression. In addition, patients receive an information booklet about depression and a community resource list.
  Arms: 2

SUMMARY:
This study will determine ways to make depression care more responsive to the needs of consumers in primary care clinics serving low-income Latinos.

DETAILED DESCRIPTION:
Depression is a serious illness that is difficult to diagnose and treat, especially in populations that underutilize mental health services. The Latino population is one such group. Accommodating patient preferences for care, provider capacities, and administrator priorities is essential to the development of effective depression care interventions that are sustainable in public sector systems. However, little is understood regarding the depression treatment preferences of low-income Latinos who have not received quality depression care and who may not feel that they can voice their opinions about their health care. In addition, little is known about the preferences, capabilities, and priorities of providers and administrators in primary care clinics. This study will determine ways to make depression care more responsive to the needs of consumers in primary care clinics serving low-income Latinos. The study will also evaluate the effectiveness of various treatments in reducing depression.

Following baseline assessments of depression treatment preferences and resources, participants in this open label study will be randomly assigned to receive collaborative care either immediately or after a waiting period. Individuals assigned to receive immediate care will undergo treatment for 12 weeks. Other participants will receive treatment at a later time. All participants will have the option to receive one of the following treatments: (1) medication management from the Depression Care Specialist (DCS) and antidepressant medication from their primary care provider (PCP); (2) cognitive-behavioral therapy from the DCS; or (3) a combination of both treatments. Depression treatment outcomes and preferences will be measured post-intervention. Provider and administrator preferences will also be measured post-intervention and potential strategies for implementing patient-centered depression care programs will be identified.

ELIGIBILITY:
Inclusion Criteria:

For Participating Patients:

* Attending one of the study clinics for primary care
* English or Spanish-speaking
* Screens positive for major depressive disorder or dysthymia

For Providers:

* All primary care providers providing at least one day of services at one of the study clinics

For Administrators:

* Administrative, medical, and nursing directors from each study site and directors of affiliated local mental health clinics

Exclusion Criteria:

For Participating Patients:

* Acutely suicidal
* Screens positive for bipolar disorder, psychotic disorder, or cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 432 (Actual)
Dates: Start 2005-11; Primary Completion 2007-10 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Depression treatment preferences as measured by a conjoint analysis survey and qualitative interviews | Measured at Week 16

SECONDARY OUTCOMES:
Depression outcomes as measured by the Patient Health Questionnaire-9 | Measured at Week 16

CONTACTS AND LOCATIONS:
Overall Officials: Isabel T. Lagomasino, MD, MSHS, Principal Investigator — University of Southern California; Megan Dwight-Johnson, MD, MPH, Principal Investigator — VA Medical Center-West Los Angeles
Locations (3):
- United States (3):
  - H. Claude Hudson Comprehensive Health Center, Los Angeles, California
  - USC Family Practice Center at California Hospital, Los Angeles, California
  - LAC+USC Outpatient Department, Los Angeles, California

REFERENCES:
- [Result] Dwight-Johnson M, Lagomasino IT, Hay J, Zhang L, Tang L, Green JM, Duan N. Effectiveness of collaborative care in addressing depression treatment preferences among low-income Latinos. Psychiatr Serv. 2010 Nov;61(11):1112-8. doi: 10.1176/ps.2010.61.11.1112. PMID 21041350